CLINICAL TRIAL: NCT01358448
Title: A Pilot Study of the Efficacy and Program Cost-effectiveness of Prevention Plus for Childhood Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UT8433B
Record Dates: First submitted 2011-05-17; First posted 2011-05-23 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Obesity
Keywords: Treatment of childhood obesity
MeSH Terms: conditions — Obesity

ARMS (3):
- Newsletter (No Intervention)
- Growth Monitoring (Experimental)
  Interventions: Behavioral: growth monitoring
- Growth Monitoring plus Family-based Behavioral Counseling (Experimental)
  Interventions: Behavioral: Growth Monitoring plus Family-based Behavioral Counseling

INTERVENTIONS:
Behavioral: growth monitoring — Caretakers will be encouraged to monitor child growth monthly.
  Arms: Growth Monitoring
Behavioral: Growth Monitoring plus Family-based Behavioral Counseling — Caretakers will monitor growth monthly in addition participating in family-based behavioral counseling
  Arms: Growth Monitoring plus Family-based Behavioral Counseling

SUMMARY:
In 2007 the Expert Committee published recommendations on the prevention and treatment of childhood obesity. These recommendations outlined four interventions intended for advancement based on the child's age, body mass index (BMI), and response to treatment. The initial stage, Prevention Plus, is to be implemented in the primary care setting and focuses on primary care providers monitoring growth monthly and delivering intervention messages that target dietary and leisure-time behaviors that most contribute to energy imbalance in children. Little research has evaluated the efficacy of these recommendations. Thus the primary goal of the proposed pilot study is to test the feasibility of the Prevention Plus stage for treating childhood overweight and obesity in a primary care setting. As the cost of interventions is a large barrier to the translation of evidence-based research into primary care settings, a second goal of the project is to evaluate program cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* between 4 to 8 years of age at the start of the intervention
* overweight or obese (≥85th BMI-for-age percentile)
* have no medical conditions that effect growth, intake or physical activity (e.g., Prader Willi Syndrome, type 2 diabetes, etc.)
* not currently participating in a weight loss program and/or taking weight loss medication
* have a primary caretaker willing to participate in the research study, receive monthly newsletters and be randomized to one of the three conditions
* caretaker must be able to read, speak and understand English and the child speak English
* have transportation to their child's primary care provider office
* family does not plan to move out of the area before March 2012

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Weight Status | Baseline and 6-month
  BMI z-score
Dietary Intake | baseline and 6-months
  dietary intake (sweetened beverages, fruits and vegetables, energy, and percent energy from fat)
Leisure-time Behaviors | Baseline and 6-months
  leisure-time behaviors (moderate-intense physical activity and television viewing)
Caretaker Feeding Behaviors | Baseline and 6-months
  Caretaker feeding behaviors (authoritative, authoritarian, permissive, restrictive) assessed by questionnaires

SECONDARY OUTCOMES:
Cost Effectiveness | 6-months
  The total program cost per 0.1 change in BMI z-score

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Knoxville Pediatric Associates, Knoxville, Tennessee
  - Healthy Eating and Activity Laboratory, Knoxville, Tennessee